CLINICAL TRIAL: NCT03881527
Title: Transaortic Native Valve Resection Using a Novel Nitinol Blade Device Rather Than a Classical Surgical Blade (Nitinol Circular Blade)
Brief Title: Nitinol Circular Blade
Acronym: NCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/14OCT/513
Record Dates: First submitted 2015-10-07; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection of the aortic valve leaflets with device (Experimental): Patients in which the aortic valve has been resected using the nitinol blade
  Interventions: Device: Aortic valve replacement using a nitinol blade
- Resection of the aortic valve leaflets in standard fashion (Other): Patients in which the aortic valve has been resected using a conventional blade or scissor
  Interventions: Procedure: aortic valve replacement

INTERVENTIONS:
Device: Aortic valve replacement using a nitinol blade — A circular nitinol blade will be inserted by to cut the aortic valve leaflets during conventional aortic valve replacement procedure
  Arms: Resection of the aortic valve leaflets with device
Procedure: aortic valve replacement — Aortic valve replacement in a standard fashion
  Arms: Resection of the aortic valve leaflets in standard fashion

SUMMARY:
The Nitinol Circular Blade (NCB) is indicated for use in patients with symptomatic aortic stenosis requiring aortic valve replacement, who are going to be operated by conventional sternotomy with native valve resection and replacement by a prosthetic aortic valve. The resection of the diseased leaflets will be performed by the NCB rather than conventional surgical blade.

DETAILED DESCRIPTION:
The patient will be under general anesthesia. The sternum will be opened fully or partially. The patient will be prepared for cardiopulmonary bypass. A transversal aortotomy will be performed as usual. The aortic valve will be exposed for the resection. The NCB will be inserted under visual control from the aorta to the left ventricle. The collection chamber will be closed and the circular blade can be advanced forward to resect the diseased native aortic valve. Once the resection is completed the device will be retrieved carefully. Complementary fine cleaning of the aortic annulus can be done by the surgeon in order to prepare the annulus to receive the prosthetic valve. After implantation of the new valve classically the aortotomy will be closed. Standard weaning of cardiopulmonary bypass will be done and the operation will be safely completed. The aim of this blade is to evaluate the resection time, test the efficiency of a circular Nitinol blade during resection of the calcified native aortic leaflets. A careful examination of the resection edges, aortic annulus, mitral valve and all surrounding tissues will be done in order to validate the efficacy of this Nitinol Circular Blade.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis defined as one or more of the following by Doppler echocardiography: mean gradient >40 mmHg; max velocity >4 m/sec; aortic valve area <=0.8 cm2.
* Symptoms related to aortic valve disease, and NYHA Functional Class II or greater
* Subject is indicated for aortic valve implantation with a biological prosthesis (tissue valve)
* Age >= 65 years
* Echocardiographically determined aortic annulus diameter >=24 mm and <=30 mm in a long-axis view
* Subject understands the implications of participating in the study and provides informed consent

Exclusion Criteria:

* Congenital unicuspid aortic valve
* Severe eccentricity of calcification, defined as calcium deposits larger than 6 mm in diameter
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Left ventricular ejection fraction <25% as determined by contrast ventriculography, or echocardiography or radionuclide angiography if contrast ventriculography not available
* Hypertrophic obstructive cardiomyopathy
* Subjects with life expectancy less than 12 months due to an underlying non-cardiac co-morbid disease
* Known hypersensitivity or contraindication that cannot be adequately controlled with pre-medication to any study medication or material, such as contrast medium or Nitinol
* Blood dyscrasia such as acute anemia, leucopenia, or thrombocytopenia; bleeding diathesis, or coagulopathy
* Renal insufficiency assessed by creatinine >2.5 mg/dl and/or end stage renal disease requiring chronic dialysis
* Poor lung function that in the investigator's opinion is prohibitive for thoracotomy
* Active peptic ulcer or GI bleeding within 3 months from the planned index procedure
* Cardiogenic shock, suspected cardiogenic shock, or hemodynamic instability requiring inotropic support or mechanical heart assistance
* Peripheral vascular disease, including abdominal and thoracic aortic disease, that could pose a problem for eventual transarterial mechanical support (e.g. intraaortic balloon pump)
* History of myocardial infarction in the last 6 weeks
* History of TIA or CVA in the last 6 months
* Subject refuses to have a blood transfusion
* Subject is currently enrolled in another investigational device or drug trial that may influence the outcome of this trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Procedural success of the resection | Hospital discharge : in average 1 week
  Resection of the aortic valve leaflets by the circular nitinol blade

SECONDARY OUTCOMES:
Complication due to the use of the device | 1 year
  Any complication related to the use of the nitinol blade

CONTACTS AND LOCATIONS:
Overall Officials: Parla ASTARCI, Md PhD, Principal Investigator — Cliniques universiatires St Luc
Locations (1):
- Parla ASTARCI, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Astarci P, Glineur D, Kefer J, Renkin J, Vanoverschelde JL, El Khoury G. "Ring pledget": a new concept for secure apex closure during transapical aortic valve implantation. Innovations (Phila). 2010 Mar;5(2):136-7. doi: 10.1097/IMI.0b013e3181cbb364. PMID 22437365
- [Result] Astarci P, Glineur D, Kefer J, D'Hoore W, Renkin J, Vanoverschelde JL, El Khoury G, Grandin C. Magnetic resonance imaging evaluation of cerebral embolization during percutaneous aortic valve implantation: comparison of transfemoral and trans-apical approaches using Edwards Sapiens valve. Eur J Cardiothorac Surg. 2011 Aug;40(2):475-9. doi: 10.1016/j.ejcts.2010.11.070. Epub 2011 Jan 20. PMID 21256045
- [Result] Astarci P, Desiron Q, Glineur D, El Khoury G. Transapical explantation of an embolized transcatheter valve. Interact Cardiovasc Thorac Surg. 2011 Jul;13(1):1-2. doi: 10.1510/icvts.2011.267757. Epub 2011 Apr 11. PMID 21486757
- [Result] Astarci P, Glineur D, Elkhoury G, Raucent B. A novel device for endovascular native aortic valve resection for transapical transcatheter aortic valve implantation. Interact Cardiovasc Thorac Surg. 2012 Apr;14(4):378-80. doi: 10.1093/icvts/ivr125. Epub 2012 Jan 9. PMID 22235001
- [Result] Astarci P, Price J, Glineur D, D'Hoore W, Kefer J, Elkhoury G, Grandin C, Vanoverschelde JL. Cerebral embolization during percutaneous valve implantation does not occur during balloon inflation valvuloplasty: prospective diffusion-weighted brain MRI study. J Heart Valve Dis. 2013 Jan;22(1):79-84. PMID 23610993
- [Result] Astarci P, Glineur D, De Kerchove L, El Khoury G. Transcatheter valve used in a bailout technique during complicated open mitral valve surgery. Interact Cardiovasc Thorac Surg. 2013 Oct;17(4):745-7. doi: 10.1093/icvts/ivt249. Epub 2013 Jun 28. PMID 23814136
- [Result] Astarci P, Etienne PY, Raucent B, Bollen X, Tranduy K, Glineur D, Dekerchove L, Noirhomme P, Elkhoury G. Transcatheter resection of the native aortic valve prior to endovalve implantation - A rational approach to reduce TAVI-induced complications. Ann Cardiothorac Surg. 2012 Jul;1(2):224-30. doi: 10.3978/j.issn.2225-319X.2012.06.15. No abstract available. PMID 23977499
- [Result] Nuis RJ, Sinning JM, Rodes-Cabau J, Gotzmann M, van Garsse L, Kefer J, Bosmans J, Yong G, Dager AE, Revilla-Orodea A, Urena M, Nickenig G, Werner N, Maessen J, Astarci P, Perez S, Benitez LM, Amat-Santos IJ, Lopez J, Dumont E, van Mieghem N, van Gelder T, van Domburg RT, de Jaegere PP. Prevalence, factors associated with, and prognostic effects of preoperative anemia on short- and long-term mortality in patients undergoing transcatheter aortic valve implantation. Circ Cardiovasc Interv. 2013 Dec;6(6):625-34. doi: 10.1161/CIRCINTERVENTIONS.113.000409. Epub 2013 Nov 26. PMID 24280965
- [Result] Gauthier C, Astarci P, Baele P, Matta A, Kahn D, Kefer J, Momeni M. Mid-term survival after transcatheter aortic valve implantation: Results with respect to the anesthetic management and to the access route (transfemoral versus transapical). Ann Card Anaesth. 2015 Jul-Sep;18(3):343-51. doi: 10.4103/0971-9784.159804. PMID 26139739
- [Result] Navarra E, Mosala Nezhad Z, Bollen X, Gielen CE, Mastrobuoni S, De Kerchove L, Raucent B, Astarci P. Endovascular resection of the native aortic valve before transcatheter aortic valve implantation: state of the art and review. Eur J Cardiothorac Surg. 2016 Sep;50(3):406-10. doi: 10.1093/ejcts/ezw027. Epub 2016 Mar 31. PMID 27032472